CLINICAL TRIAL: NCT04122794
Title: The Role of Unsteady Wall Shears Stress Stimuli on Human Umbilical Vein Endothelial Cells (HUVECs) Harvested From Umbilical Cords
Brief Title: The Role of Unsteady Wall Shears Stress Stimuli on Human Umbilical Vein Endothelial Cells Harvested From Umbilical Cords
Acronym: HUVEC
Status: Terminated | Type: Observational
Why Stopped: Impact of Covid-19 and staffing has required us to suspend this study
Sponsor: University Hospital of Limerick (Other)
Collaborators: University of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Professor Eamon Kavanagh Prinicipal Investigator, University Hospital of Limerick
Other Study IDs: DVS006
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Vascular Diseases
Keywords: Endothelial Cells
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Endothelial cells will be retrieved from the endothelial vein of human umbilical cord tissue that would be otherwise discarded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to obtain and test endothelial cells (EC's) from umbilical cords to examine specific properties of these cells which make up the inner lining of blood vessels.

DETAILED DESCRIPTION:
Mechanical testing will be performed on the Ec's to see how the cells reacts and ultimately how the blood vessel is affected.

A central role in the mechanism that defines the nature of vessel remodelling is played by endothelial cells. EC's are extremely sensitive to the frictional forces exerted on a unit of the endothelial area by blood flow. This mechanical stimulus is known as wall shear stress (WSS). WSS experienced by EC's in-vivo is unsteady due to the unsteady nature of blood flow produced during the cardiac cycle and due to the complex nature of the vascular tree.

The extent to which this applies to venous cells and tissue remains unknown and it is the focus of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are attending the Maternity Services who are pregnant and due for routine delivery.
* Aged 18- 40 years.
* Are willing and capable to voluntarily sign a statement of informed consent to take part in this investigation.
* Patients due to give birth to twins will be included in this study. Women having both "normal" delivery and caesarean section delivery will be included in this study.

Exclusion Criteria:

* Patients unable to provide informed consent.
* Patients who are under the age of 18 and over the age of 40 years.
* Patients who are deemed unsuitable due to any circumstances as deemed appropriate by the Consultant.
* Patients with a Blood Borne Virus (HIV Type 1, HIV Type 2, Hepatitis B, Hepatitis C) will be excluded from the study.
* Patients with diabetes that is not gestational in nature will be excluded from this study.
* Patients due to deliver triplets or more will be excluded from this study.
* Patients who deliver their baby before 37 weeks gestation will not have umbilical cord tissue retained for study purposes.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Women attending Maternity Services in Limerick who are pregnant and due for routine delivery that meet all the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
The identification of Endothelial Cell phenotype | 2 years
  To identify this phenotype by assessing the endothelial identity markers, the endothelial to mesenchymal transition markers and the regulation of genes involved in EC quiescence.

CONTACTS AND LOCATIONS:
Overall Officials: Eamon Kavanagh, MD FRCSI, Principal Investigator — University Hospital of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No